CLINICAL TRIAL: NCT02396199
Title: Zenith® p-Branch® Pivotal Study
Brief Title: Zenith® p-Branch® Endovascular Graft Pivotal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-09
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Aortic Aneurysm Abdominal
Keywords: Abdominal aortic aneurysm; Endovascular; Juxtarenal; Pararenal; Fenestrated
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Endovascular (Experimental): Endovascular treatment using the Zenith® p-Branch® in combination with the Atrium iCAST™ covered stents
  Interventions: Device: Zenith® p-Branch® in combination with the Atrium iCAST™ covered stents

INTERVENTIONS:
Device: Zenith® p-Branch® in combination with the Atrium iCAST™ covered stents — Instead of making a large incision in the abdomen, the physician makes a small incision near each hip to insert, and guides the study device(s) into place in the aorta.
  Other Names: Endovascular graft; Endovascular stent; Stent-graft; Fenestrated graft

SUMMARY:
The Zenith® p-Branch® Pivotal Study is a clinical trial approved by FDA to study the safety and effectiveness of the Zenith® p-Branch® endovascular graft in combination with the Atrium iCAST™ covered stents in the treatment of abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Pararenal or juxtarenal AAA ≥5.0 cm in diameter or 2 times the normal aortic diameter
* Pararenal or juxtarenal AAA with history of growth ≥0.5 cm/year
* Saccular aneurysm with aortic diameter greater than 1.5 times the normal aortic diameter that is deemed to be at risk for rupture based upon physician interpretation

Exclusion Criteria:

* Age <18 years
* Life expectancy <2 years
* Pregnant, breast-feeding, or planning on becoming pregnant within 60 months
* Inability or refusal to give informed consent by the patient or a legally authorized representative
* Unwilling or unable to comply with the follow-up schedule
* Simultaneously participating in another investigative device or drug study. (The patient must have completed the primary endpoint of any previous study at least 30 days prior to enrollment in this study.)
* Additional medical restrictions as specified in the Clinical Investigation Plan
* Additional anatomical restrictions as specified in the Clinical Investigation Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2021-04-01 (Actual); Study Completion 2025-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Farber, MD, Principal Investigator — University of North Carolina
Locations (27):
- United States (27):
  - University of Alabama Birmingham Hosptial, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center-Dignity Health, Phoenix, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente, San Francisco, California
  - Stanford University Medical School, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Boca Raton Community Hospita, Boca Raton, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Minneapolis Heart Inst. Foundation, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Barnes Jewish Hospital Plaza, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - New York University - Langone Medical Center, New York, New York
  - Mount Sinai Roosevelt, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital - Smith Tower, Houston, Texas
  - Baylor Scott and White Research Institute, Irving, Texas
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endovascular
Started | 80
Started 6-Month | 79
Completed 6-Month | 76
Started 12-Month | 76
Completed | 75
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One participant had an unreported race/ethnicity
  Participants
    Black(origins of Africa): number analyzed (Participants) | 79
    Black(origins of Africa) | 7
    White(origins of Europe, Middle East, or North Africa): number analyzed (Participants) | 79
    White(origins of Europe, Middle East, or North Africa) | 72

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success Proportion
Description: Technical success and freedom from type 1 and type 3 endoleaks which require intervention, aneurysm growth, related SAE's, and related major complications
Time Frame: 12 months
Population: Eight patients had incomplete outcome data either due to death, loss to follow-up, missed visits, or any combination thereof.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Endovascular
Number analyzed (Participants) | 72
Proportion of participants | 0.917 [0.827 to 0.969]
Statistical Analysis 1: Comparison: Endovascular; Test type: Superiority; p = 0.006, Fisher Exact — One-sided test; Proportion of participants = 0.917, 95% CI 1-sided [lower limit 0.827] — Exact test, One-sided 95%, with lower limit (0.827)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Endovascular: Endovascular treatment using the Zenith® p-Branch® in combination with the Atrium iCAST™ covered stents
  Zenith® p-Branch® in combination with the Atrium iCAST™ covered stents: Instead of making a large incision in the abdomen, the physician makes a small incision near each hip to insert and guide the study device(s) into place in the aorta.
Arm/Group | Endovascular
All-Cause Mortality (participants affected / at risk) | 4/80
Serious Adverse Events (participants affected / at risk) | 25/80
Other Adverse Events (participants affected / at risk) | 8/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=80)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 3 (3)
Vascular stent occlusion (General disorders) | 6 (7)
Vascular stent stenosis (General disorders) | 2 (2)
Vascular stent thrombosis (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 2 (3)
Renal mass (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Debridement (Surgical and medical procedures) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=80)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Stent-graft endoleak (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT02396199/Prot_SAP_000.pdf